CLINICAL TRIAL: NCT07342348
Title: Using Power Mobility Training to Promote Arm & Hand Function in Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grand Valley State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26-065-H
Record Dates: First submitted 2026-01-08; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy; Hemiplegia, Infantile
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm- and hand-use focused power mobility training group (Experimental): These arm- and hand-use focused power mobility training activities will be provided via a ride-on toy and will encompass both navigational/maneuvering activities and play-based reaching and grasping activities embedded into the navigational/maneuvering activities. During power mobility training activities, children will be asked to wear a soft mitten or sock on their preferred hand to help them remember to use their less preferred hand and arm.
  Interventions: Other: Arm- and hand-use focused power mobility training

INTERVENTIONS:
Other: Arm- and hand-use focused power mobility training — These arm- and hand-use focused power mobility training activities will encompass both navigational/maneuvering activities and play-based reaching and grasping activities embedded into the navigational/maneuvering activities. During power mobility training activities, children will be asked to wear a soft mitten or sock on their preferred hand to help them remember to use their less preferred hand and arm.

SUMMARY:
Approximately 40% of children with ambulatory cerebral palsy have significant functional asymmetries in arm and hand function. Children with these significant functional asymmetries have difficulties using their more-affected (less preferred) arm and hand in daily activities, especially true in daily activities requiring bilateral hand and arm use. Recent research suggests that power mobility training provided via a ride-on toy may help to motivate these children to use their less preferred arm and hand. This research further notes that participation in power mobility training designed to encourage a child to use their less preferred arm and hand also may help to improve their arm and hand function and use in their daily activities. This exploratory study seeks to explore an innovative intervention using arm- and hand-use focused power mobility training activities, encompassing both navigational/maneuvering activities and embedded play-based reaching and grasping activities. During power mobility training activities, children will be asked to wear a soft mitten or sock on their preferred hand to help them remember to use their less preferred hand and arm.

The purpose of this exploratory study is to examine both the effect and feasibility of a 6-week laboratory-based arm-and hand-use focused power mobility training program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy
* Demonstrates significantly less functional use of one arm and hand
* Can get on and off the a ride-on toy with minimal assistance from the researchers
* Can maintain a sitting position on the a ride-on toy
* Has sufficient functional vision to safely maneuver the a ride-on toy
* Has their own bicycle helmet that fits them well and is in good working condition

Exclusion Criteria:

* Hand or arm surgery within the past 6 months
* Their weight exceeds device limits (more than 120 pounds)
* They do not demonstrate sufficient balance and control in sitting to safely use the ride-on toy
* If they cannot safely participate in arm- and hand-use focused power mobility training activities.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | From enrollment to the end of treatment at 6 weeks
  The Canadian Occupational Performance Measure rates parent/caregiver perceptions of their child's performance of 5 arm and hand skills. Each skill is rated from a minimum of 1 to a maximum of 10. A higher score indicates a better outcome. The total score on all 5 items ranges from a minimum of 5 to a maximum of 50. A higher score indicates a better outcome.
ABILHAND-Kids-CP Questionnaire | From enrollment to the end of treatment at 6 weeks
  The ABILHAND measures parents' perceptions of their child's manual ability and provides a comprehensive evaluation of the child's functional arm and hand ability. Parents estimate their child's ease or difficulty in performing 17 activities. Each activity is rated using a 3-point Likery scale as follows: 'Impossible=0, Difficult=1, Easy=2. Higher scores indicate a better outcome.

SECONDARY OUTCOMES:
Shriner's Hospital Upper Extremity Evaluation | From enrollment to the end of treatment at 6 weeks
  The Shriner's Hospital Upper Extremity Evaluationis a 16-item video-recorded test to assess spontaneous use and dynamic alignment of the affected UE during bimanual tasks. Higher scores indicate better outcomes.
Grip strength | From enrollment to the end of treatment at 8 weeks
  Children's grip strength will be measured bilaterally. Higher values indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa K. Kenyon, PT, DPT, PhD, PCS, Principal Investigator — Grand Valley State University
Locations (1):
- Grand Valley State University, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Srinivasan SM, Kataria K, Yorns W Jr, Moore TE, Yoo C, Kumavor PD, Morgan K, Friel K. A novel program including ride-on toys to improve upper extremity function in children with hemiplegia: a randomized controlled trial. Disabil Rehabil Assist Technol. 2026 Jan;21(1):173-186. doi: 10.1080/17483107.2025.2534436. Epub 2025 Jul 21. PMID 40689868
- [Background] Srinivasan S, Shahane V, Kumavor P, Morgan K, Friel K. Joystick-Operated Ride-On Toys as a Therapy Adjunct for a Child With Hemiplegia: A Case Report. Pediatr Phys Ther. 2025 Jul 1;37(3):371-379. doi: 10.1097/PEP.0000000000001209. Epub 2025 Jun 27. PMID 40587602
- [Background] Amonkar N, Kumavor P, Morgan K, Bubela D, Srinivasan S. Feasibility of Using Joystick-Operated Ride-on-Toys to Promote Upper Extremity Function in Children With Cerebral Palsy: A Pilot Study. Pediatr Phys Ther. 2022 Oct 1;34(4):508-517. doi: 10.1097/PEP.0000000000000944. Epub 2022 Aug 30. PMID 36044637